CLINICAL TRIAL: NCT03210792
Title: Comparison of the Effectiveness in Pain Reduction Between a Rib Splint Produced in the ER and a Manufactured Rib Splint: Preliminary Clinical Study
Brief Title: Comparison Manufactured Rib Splint With Hand-made Rib Splint
Acronym: CMRSHRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, LEE YOON-JE, Clinical Assistant Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIBSPLINTPRESTUDY
Record Dates: First submitted 2017-07-04; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCO Rib Splint (Active Comparator): Subjects were applied Chrisofix® Chest Orthosis (Manufactured Rib Splint) for Rib Fractures treatment.
  Interventions: Device: Application of Rib Splint
- Handmade Rib Splint (Experimental): Subjects were applied Handmade Rib Splint for Rib Fractures treatment.
  Interventions: Device: Application of Rib Splint

INTERVENTIONS:
Device: Application of Rib Splint — Investigators randomly apply handmade Rib Splint or manufactured Rib Splint to subjects.

SUMMARY:
A pilot study for a prospective randomized clinical trial was conducted to compare subjects using the CCO (Group-A) with those using the ER-splint (Group-B) before and after the intervention.

The primary outcome was difference in the level of pain based on the visual analogue scale (VAS) between before and after intervention in each group during forceful and resting respiration.

VAS : Visual analogue scale CCO : Chrisofix® Chest Orthosis

DETAILED DESCRIPTION:
Investigators performed VAS assessments to determine the level of pain in the subjects with RFs during resting and forceful respiration. Investigators applied either the CCO rib splint or the ER splint to the RF subjects in a randomized order. At 30 minutes after splint application, investigators repeated the VAS assessments during resting and forceful respiration. Subsequently, additional pain control was provided via intravascular drug injection.

RF : Rib fractures VAS : Visual analogue scale CCO : Chrisofix® Chest Orthosis

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have rib fractures and age was over 18 years old

Exclusion Criteria:

* Investigators excluded subjects with cardiopulmonary dysfunction, poly-trauma, flail chest, damage to an internal organ, or alcoholism and subjects who did not consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-07-10 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of each intervention based on the VAS scores in each group during resting and forceful respiration | We check a pain scale at 30 minutes after splint application
  Comparison CCO Rib splint with Handmade Rib splint about pain reduction